CLINICAL TRIAL: NCT00044109
Title: Static Magnets In The Treatment of Sciatica
Brief Title: Magnets in the Treatment of Sciatica
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020274; 02-D-0274
Record Dates: First submitted 2002-08-17; First posted 2002-08-19 (Estimated); Last update posted 2006-06-26 (Estimated); Status verified 2006-06

CONDITIONS: Low Back Pain; Sciatica
Keywords: Pain; Low Back; Radiculopathy; Electromagnetic Treatment; Back Device; Sciatica; Low Back Pain
MeSH Terms: conditions — Low Back Pain; Sciatica; Pain; Radiculopathy

INTERVENTIONS:
Device: Magnets

SUMMARY:
Despite much popularity among the public, magnetic devices used for the treatment of various musculoskeletal and neuropathic pain syndromes have been the subject of few randomized controlled trials.

We propose to study the effects of permanent 200 gauss magnets on lumbar radicular pain. This study will include 52 men and women of all ethnic backgrounds between the ages of 28 and 75 who have had signs and symptoms of sciatica for 3 months or more.

This is a double-blind, randomized, placebo-control, two phase study. In the first phase, after one week baseline, subjects will be randomized to 4 different treatments in a cross-over design. These 4 treatments which will last two weeks each are: 1 magnetic device positioned in 2 different ways along the spinal axis (up-down along the lumbo-sacral spine and left-right across the lumbo-sacral spine), a sham device of similar configuration and a no treatment control. The length of phase I will be 8 weeks. At the end of this phase, codes will be broken to select the magnetic device associated with the greatest amount of pain score reduction. During the second phase which will also be double-blinded, subjects will be randomized to wear the selected magnetic device and sham in a cross-over design. Each of the 2 periods will be 5 weeks in duration. The primary outcome measures will be the daily pain score in the leg. Daily pain level in the low back and the back and leg combined in addition to the patients' quality of life and activities of daily living will be secondary outcome measures as assessed by the SF 36, Oswestry, and Beck depression inventory.

DETAILED DESCRIPTION:
Despite much popularity among the public, magnetic devices used for the treatment of various musculoskeletal and neuropathic pain syndromes have been the subject of few randomized controlled trials.

We propose to study the effects of permanent 200 gauss magnets on lumbar radicular pain. This study will include 52 men and women of all ethnic backgrounds between the ages of 28 and 75 who have had signs and symptoms of sciatica for 3 months or more.

This is a double-blind, randomized, placebo-control, two phase study. In the first phase, after one week baseline, subjects will be randomized to 4 different treatments in a cross-over design. These 4 treatments which will last two weeks each are: 1 magnetic device positioned in 2 different ways along the spinal axis (up-down along the lumbo-sacral spine and left-right across the lumbo-sacral spine), a sham device of similar configuration and a no treatment control. The length of phase I will be 8 weeks. At the end of this phase, codes will be broken to select the magnetic device associated with the greatest amount of pain score reduction. During the second phase which will also be double-blinded, subjects will be randomized to wear the selected magnetic device and sham in a cross-over design. Each of the 2 periods will be 5 weeks in duration. The primary outcome measures will be the daily pain score in the leg. Daily pain level in the low back and the back and leg combined in addition to the patients' quality of life and activities of daily living will be secondary outcome measures as assessed by the SF 36, Oswestry, and Beck depression inventory.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Low back pain of 3 months duration or longer present at least 5 out of 7 days a week
  2. Age between 28-80 at the start of the study
  3. Men and women of all ethnicities
  4. Signs and symptoms of lumbar radiculopathy. In this study chronic lumbar radicular signs and symptoms are defined as pain located in the lower lumbar spine corresponding to L1 and below for at least 3 months with radicular characteristics, i.e. pain described as sharp, burning, with numbness and/or tingling.
  5. Ability to understand the study measures and mentally capable to give consent to participate in the study (based on an 8th grade education level)
  6. Willingness to refrain from making changes in non-study medications taken for sciatica
  7. Patients with failed back syndrome.
  8. Pain level of at least 4/10 on average on a scale of 0 to 10 for the past month
  9. Pain not attributable to malignancy, inflammatory arthritis such as rheumatoid arthritis, or infection by previous examinations or by laboratory testing
  10. Patients' agreement to keeping a log of their pain level and documentation of compliance with wearing of back device.
  11. Patients' agreement not to make changes in pain medication type of dosing during the study.
  12. Women of reproductive age agreeing to undergo a pregnancy test at baseline.

EXCLUSION CRITERIA:

1. Patients with pacemakers
2. Patients with mechanical heart pumps
3. Pregnancy or breast feeding
4. Presence of pain of greater intensity in any other location than the low back or the leg
5. History of fibromyalgia as described by Wolfe F et al. (1990) (a minimum of 11 out of 18 points of tenderness must be present to satisfy criteria for fibromyalgia)
6. History of spinal unstability (as defined by X-ray, CT scan or MRI of grade II spondylolisthesis or greater)
7. Cognitive impairment such that the individual is unable to give informed consent, complete study data collection tools or required study visits
8. Unwillingness to use adequate contraception excluding oral contraceptive medications (such as barrier methods with spermicide simultaneously) for women
9. Presence of other medical condition presenting with numbness and pain in lower extremities, such as diabetic polyneuropathy and peripheral vascular disease
10. History of inflammation arthritis (rheumatoid arthritis, SLE)
11. Presence of active cancer
12. History of spinal infection
13. Patients s/p spinal fusion with spinal rods over the lower lumbar spine

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2002-08; Study Completion 2006-06

PRIMARY OUTCOMES:
Daily overall pain level, pain in the low back and pain in the lower extremities will be rated on a scale of 0 to 10.

SECONDARY OUTCOMES:
Baseline and end of period 1 and 2 of Phase II: Pain symptoms, Pain level with walking, Use of pain meds, Use of other non-medication treatments, questionnaire: SF 36, Oswestry and Beck Depression, Days of disability. End of Study: Patient preference.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Blank M, Soo L. Optimal frequencies for magnetic acceleration of cytochrome oxidase and Na,K-ATPase reactions. Bioelectrochemistry. 2001 Mar;53(2):171-4. doi: 10.1016/s0302-4598(00)00128-8. PMID 11339304